CLINICAL TRIAL: NCT04642807
Title: Management of Type 1 Supracondylar Humeral Fractures: a Multicentre Randomized Control Trial
Brief Title: Management of Type 1 Supracondylar Humeral Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Queensland Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Anthony Cooper, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-02942
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Elbow Fracture; Trauma
Keywords: Supracondylar humeral fracture; Pediatric elbow fracture
MeSH Terms: conditions — Elbow Fractures; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 "Long-arm full cast and routine follow-up" (Active Comparator): Patients assigned to Group 1 will be placed in a long arm cast, at 90-100 degrees in neutral rotation. A referral will then be made to the orthopedic department and the patient reviewed at week 3 with cast removal, clinical assessment and radiographic assessment as determined by the normal practice at the local center.
  Interventions: Procedure: Long arm full cast
- Group 2 "Long-arm soft cast and no clinical or radiographic follow-up" (Experimental): Patients assigned to group 2 will be placed in a long arm cast at 90-100 degrees in neutral rotation. They will be given verbal and written information on the injury, when and how to remove the cast and contact details if there are any concerns.
  Since they will not be attending clinical follow-up, an email or telephone survey will be undertaken at 3 weeks and after 6 months. The survey will inquire initially about pain, unplanned returns to the Family Physician and hospital, complications, parent/patient satisfaction and a standardized patient reported outcome score will be taken. Please see attached documentation for the itemized survey questions. The 6 month follow-up will include photographs and an illustrated guide will be given to the families on how to obtain pictures of maximal flexion, extension and the child's carrying angle (attached). Measurements of range of motion from photographs are considered comparable to clinical assessment of range of motion
  Interventions: Procedure: Long arm soft cast

INTERVENTIONS:
Procedure: Long arm soft cast — Participants in group 2 will have a long arm soft cast applied without clinical or radiological follow up.
  Arms: Group 2 "Long-arm soft cast and no clinical or radiographic follow-up"
Procedure: Long arm full cast — Participants in group 1 will have a long arm full cast applied.
  Arms: Group 1 "Long-arm full cast and routine follow-up"

SUMMARY:
This study compares the clinical outcomes of treating pediatric Type 1 supracondylar fracture with a long arm soft cast and no clinical or radiographic follow-up versus the standard treatment in a long arm cast with clinical follow-up.

This is the first multicenter randomized control trial looking at the clinical effectiveness, safety and parental satisfaction of managing inherently stable Type I supracondylar fractures without clinical or radiological follow-up. If found to be safe; children can be managed effectively without in-person follow-up, freeing clinic appointments to children on the waiting list and in these COVID times avoiding unnecessary contacts.

DETAILED DESCRIPTION:
PURPOSE The purpose of this study is to compare the clinical outcomes and parental satisfaction of treating pediatric Type I supracondylar fractures with a long arm soft cast and no clinical or radiographic follow-up versus standard treatment in a long arm cast with clinical follow-up.

HYPOTHESIS We propose that with clear instructions given to parents in the form of a clinical consultation at soft cast application and written instructions, a Type I supracondylar fracture can be managed with no significant change in pain, without formal in-person clinic consultation, that the treatment will proceed without any negative consequences and the treatment will be met with high parent satisfaction.

JUSTIFICATION The limiting of unnecessary patient visits, X-rays and interactions has taken on a new importance with the ongoing COVID-19 pandemic. Any research that can limit unnecessary risk to our patients, parents and families in terms of contacts should be considered and implemented now more than ever.

OBJECTIVES Our objective is to determine whether Type I supracondylar fractures can be managed safely and effectively without clinical and radiographic follow-up x-rays.

With the COVID-19 pandemic, there has been an increased need to minimize patient interactions for the safety of patients and healthcare workers alike. Typically, these fractures can be managed with minimal intervention. A cast is applied primarily to alleviate pain and the child is required to return to the hospital to have the cast removed.

A soft cast provides adequate immobilization of the fracture but can be removed at home by parents. If this can be shown to provide equivalent pain relief and a similar safety profile then there will be clear benefits at this time in limiting in-person visits and thus potential COVID-19 contacts. In a non-COVID-19 period, there will also be secondary health economic benefits by reducing out-patient follow-up visits.

If our study proves there are no negative consequences then this treatment regime could be simply and rapidly implemented at centers around the world. Additionally if successful it could also be potentially applied to the management of other undisplaced and stable fractures, which would have a considerable impact on the interactions and unnecessary contacts.

RESEARCH DESIGN This study is a prospective multicenter randomized control trial evaluating patients treated with a consistent protocol assessing clinical effectiveness, safety and parental satisfaction with the management of Type I supracondylar fractures with a period of casting and no in-person clinical or radiographic follow-up compared to cast and routine follow-up (standard current practice).

STATISTICAL ANALYSIS All baseline and relevant center and demographic information will be summarized between trial arms via appropriate summary statistics (medians and IQRs for continuous variables and counts for categorical variables).

The primary outcome and any other continuous outcomes will be assessed with a mixed effects model with a random intercept for study center, and a single covariate for treatment group. The coefficient from this model represents the estimated mean difference between groups and will be reported with a 95% confidence interval. Binary outcomes such as unplanned return to hospital will be analyzed similarly with mixed effects logistic regression and odds ratios and 95% confidence intervals will be reported.

As the objective is to show that no follow up is not inferior to standard of care, we prespecify a 20% margin of difference as clinically equivalent for the primary outcome of difference in the pain scale between groups (i.e. 2 points on 10-point scale). Therefore, if the lower bound of the 95% confidence interval from the mixed effects model lies above 20% of the mean, we will treat this as confirmation of non-inferiority. If the entire interval lies within +/- 20% this will be taken as equivalence.

Effect modification of the comparability in the primary outcome between groups will be assessed by including interaction terms with relevant baseline risk factors. Sensitivity analyses will be based on the inclusion of patient and center level covariates thought to impact the primary outcomes and multiple imputation for missing outcomes due to possible differential follow up between groups.

Analyses will be conducted using R statistical software, and a significance level of 0.05 will be used for all analyses. A formal statistical analysis plan will be finalized by all investigators prior to.

ELIGIBILITY:
Inclusion Criteria:

- Children 3 to 8 years of age with a diagnosed supracondylar humerus fracture Type 1 (undisplaced).

Exclusion Criteria:

* Children diagnosed with a Type II or III supracondylar fracture or any other elbow injury
* Children who present with neurovascular compromise associated with their fracture
* Children who have been previously diagnosed with a metabolic or structural bone disease that predisposes them to fractures

Diagnostic criteria for a Type I supracondylar fracture will include either:

A) A clear fracture line through the supracondylar region with no displacement or angulation of the distal humerus (including a normal anterior humeral line that intersects the capitellum) OR B) The absence of a clear fracture line but history of an extension injury to the arm AND tenderness at the elbow AND local swelling AND presence of a posterior fat pad on plain radiographs.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Faces Pain Scale - Revised (FPS-R) | 3 weeks post fracture
  The Faces Pain Scale - Revised (FPS-R) will be used to measure pain score. The scale uses a 0 to 10 metric that is in close linear relationship with a visual analogue pain scale. 0 is no pain and 10 is very much pain.

SECONDARY OUTCOMES:
Number of unplanned visits to the hospital or family physician | During cast treatment
  Any visits to the hospital or family physician that were not planned
Is parental satisfaction higher when they are empowered to remove a splint at home and follow a physician directed treatment program? | 3 Weeks post fracture
Is there a difference in range of elbow joint motion between the two groups at 6 months post fracture? | 6 months post fracture
• Is the difference in carrying angle from the contralateral arm at 6 months post fracture similar in children undergoing no clinical follow up or radiographic follow up compared to children undergoing routine follow-up as per the standard of care? | 6 months post fracture

CONTACTS AND LOCATIONS:
Locations (2):
- Queensland Children's Hospital, 501 Stanley Street,, South Brisbane, Australia
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva M, Sadlik G, Avoian T, Ebramzadeh E. A Removable Long-arm Soft Cast to Treat Nondisplaced Pediatric Elbow Fractures: A Randomized, Controlled Trial. J Pediatr Orthop. 2018 Apr;38(4):223-229. doi: 10.1097/BPO.0000000000000802. PMID 29517983
- [Background] Witney-Lagen C, Smith C, Walsh G. Soft cast versus rigid cast for treatment of distal radius buckle fractures in children. Injury. 2013 Apr;44(4):508-13. doi: 10.1016/j.injury.2012.11.018. Epub 2012 Dec 22. PMID 23265786
- [Background] Shrader MW. Pediatric supracondylar fractures and pediatric physeal elbow fractures. Orthop Clin North Am. 2008 Apr;39(2):163-71, v. doi: 10.1016/j.ocl.2007.12.005. PMID 18374807
- [Background] Beaty JH and Kasser JR. The Elbow Region: General Concepts in the Pediatric Patient. In: Beaty JH and Kasser JR (editors). 6th ed. Philadelphia: Lippincott, Williams & Wilkins; 2006.
- [Background] Wilkins KE and Rockwood CA. Fractures and Dislocations of the Elbow Region. 4th ed. Philadelphia: Lippincott-Raven; 1996.
- [Background] GARTLAND JJ. Management of supracondylar fractures of the humerus in children. Surg Gynecol Obstet. 1959 Aug;109(2):145-54. No abstract available. PMID 13675986
- [Background] Barton KL, Kaminsky CK, Green DW, Shean CJ, Kautz SM, Skaggs DL. Reliability of a modified Gartland classification of supracondylar humerus fractures. J Pediatr Orthop. 2001 Jan-Feb;21(1):27-30. doi: 10.1097/00004694-200101000-00007. PMID 11176349
- [Background] Skaggs DL, Mirzayan R. The posterior fat pad sign in association with occult fracture of the elbow in children. J Bone Joint Surg Am. 1999 Oct;81(10):1429-33. doi: 10.2106/00004623-199910000-00007. PMID 10535592
- [Background] Symons S, Rowsell M, Bhowal B, Dias JJ. Hospital versus home management of children with buckle fractures of the distal radius. A prospective, randomised trial. J Bone Joint Surg Br. 2001 May;83(4):556-60. doi: 10.1302/0301-620x.83b4.11211. PMID 11380131
- [Background] Meislin MA, Wagner ER, Shin AY. A Comparison of Elbow Range of Motion Measurements: Smartphone-Based Digital Photography Versus Goniometric Measurements. J Hand Surg Am. 2016 Apr;41(4):510-515.e1. doi: 10.1016/j.jhsa.2016.01.006. Epub 2016 Feb 13. PMID 26880499
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Tsze DS, Hirschfeld G, von Baeyer CL, Bulloch B, Dayan PS. Clinically significant differences in acute pain measured on self-report pain scales in children. Acad Emerg Med. 2015 Apr;22(4):415-22. doi: 10.1111/acem.12620. Epub 2015 Mar 13. PMID 25773461
- [Background] Francis Ruvuna. Unequal Center Sizes, Sample Size, and Power in Multicenter Clinical Trials. Drug Inf 2004;38:387-94.